CLINICAL TRIAL: NCT06760156
Title: Phase 2 Study of Tafasitamab and Lenalidomide as First Salvage Therapy for Residual Large B Cell Lymphoma After Axicabtagene Ciloleucel
Brief Title: Tafasitamab and Lenalidomide as First Salvage Therapy for Residual Large B Cell Lym
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21955
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Large B-cell Lymphoma
MeSH Terms: interventions — tafasitamab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tafasitamab and Lenalidomide Treatment (Experimental): Participants will receive the study drug, Tafasitamab, intravenously on a weekly basis for the first three 28-day cycles (Cycles 1-3) and then every 2 weeks starting at Cycle 4 onwards. Participants will take the study drug, Lenalidomide, once daily for 21 days out of each 28-day cycle for 6 cycles.
  Interventions: Drug: Tafasitamab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Tafasitamab — The recommended dose of tafasitamab is 12 mg/kg.
Drug: Lenalidomide — The starting dose for lenalidomide will be 25 mg PO daily.

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of tafasitamab and lenalidomide in participants with Large B Cell Lymphoma (LBCL) after axicabtagene ciloleucel (axi-cel) treatment. Participants will be asked to spend about 12 months in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented history of large B-cell lymphoma, including diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma, and DLBCL arising from follicular lymphoma.
* Adult males or females must be of age ≥18 years or older at time of signing informed consent.
* Patients must be capable of understanding the protocol with willingness to comply with all study procedures including availability for the duration of the study.
* Patients must be able to understand and willing to sign a written informed consent form (ICF) document.
* Measurable PET/CT positive disease (partial response or stable disease per the 2014 Lugano Classification) on PET/CT obtained at least 21 days after, but no more than 60 days after CAR-T with axicabtagene-ciloleucel.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Participants must have adequate organ and bone marrow function.
* Patients must have adequate hepatic function.
* Patients must have adequate renal function.
* Baseline Oxygen Saturation >92% on room air.
* Females of reproductive potential must avoid pregnancy for at least 4 weeks before beginning lenalidomide therapy, during therapy, during dose interruptions and for at least 4 weeks after completing therapy. Females must commit either to abstain continuously from heterosexual sexual intercourse or to use two methods of reliable birth control, beginning 4 weeks prior to initiating treatment with lenalidomide, during therapy, during dose interruptions and continuing for 4 weeks following discontinuation of lenalidomide therapy.

Exclusion Criteria:

* Patients who are currently receiving or who have received any investigational study agent ≤4 weeks prior to the screening visit are ineligible.
* Detectable cerebrospinal fluid malignant cells, brain metastases, or active central nervous system (CNS) lymphoma after CAR T cell administration.
* History or presence of CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
* Presence of bacterial, viral, fungal, and/or other infection of any origin that is uncontrolled and/or requires intravenous (IV) antimicrobials for treatment.
* Known cardiac atrial or cardiac ventricular lymphoma involvement.
* History of symptomatic pulmonary embolism within 6 months of enrollment.
* Known primary immunodeficiency.
* History of autoimmune disease (e.g. Crohn's disease, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.
* History of hypersensitivity, allergy or severe skin reactions to lenalidomide (e.g., angioedema, Stevens-Johnson syndrome, toxic epidermal necrolysis).
* History of hypersensitivity, allergy or previous exposure to tafasitamab.
* Any medical condition deemed by the treating physician likely to interfere with assessment of safety or efficacy of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | Up to 3 months
  Complete Response Rate (CRR) is defined as the proportion of patients with a Complete Response (CR)

SECONDARY OUTCOMES:
Objectives Response Rate (ORR) | Up to 12 months
  Defined as the incidence of either a complete response (CR) or a partial response (PR) per Lugano Classification as determined by study investigators.
Duration of Response (DoR) | Up to 12 months
  DoR is defined as the date of their first objective response to disease progression per Lugano Classification as determined by study investigators or death from any cause.
Progression Free Survival (PFS) | Up to 12 months
  Defined as the time from tafasitamab infusion date to the date of disease progression per Lugano Classification as determined by study investigators or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Locke, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States